CLINICAL TRIAL: NCT03446079
Title: Relationship of Skin Related Single Nucleotide Polymorphisms to Clinical Response to a Topical Skin Care Product
Brief Title: Relationship of Skin Related SNP to Topical Skin Care Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HelicalCodeMD (Industry)
Collaborators: 23andMe, Inc. (Industry); Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HCODE1
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Genetics; Skin Aging
Keywords: Genetic; Skin; Anti Aging; SNP
MeSH Terms: interventions — Genetic Testing

STUDY DESIGN:
Intervention Model Description: Cross sectional will utilize gene-specific candidate and genome wide association analysis to identify SNP's that may be associated with response to a topical product.
Masking Description: Investigators and participants will be blinded to the results genetic testing results during the trial duration. Only participants will be blinded to the identity of the study product.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Subjects (Experimental): Male or female subjects 21 or older that meet the specified inclusion/exclusion criteria taking genetic test and applying topical anti aging cream per the protocol.
  Interventions: Other: Topical Anti Aging Cream

INTERVENTIONS:
Other: Topical Anti Aging Cream — Primary Subjects will take a saliva based genetic test and apply a topical anti aging cream for 6 weeks.
  Other Names: Genetic Test (for association purposes only)

SUMMARY:
Demonstrate the relationship between single nucleotide polymorphisms (SNP) and response to a topical skin care product.

DETAILED DESCRIPTION:
Cross sectional study will utilize gene-specific candidate and genome wide association analysis to identify SNP's that may be associated with response to a topical product. Investigators and patients will be blinded to the genetic test results, and participants will be blinded to the skin product applied.

ELIGIBILITY:
Inclusion Criteria:

1. At least 21 years old in general good health as determined by a health questionnaire.
2. Willingness to cooperate and participate by following study requirements and to report any adverse symptoms immediately.
3. Willingness to discontinue the use of all facial products other than the assigned test material and their regular brands of glamour products. The glamour products must be the subject's regular brand and have been used for a minimum of one month prior to the start of the study.
4. Willingness to remove make up at least 30 minutes prior to each scheduled clinic visit. No other topical products should be applied to the face until the study visit has been completed.
5. Willingness to avoid daily direct sun exposure on the face, whether natural or at tanning salons.
6. Willingness to discontinue antiaging cosmetics including alpha hydroxyacid products (including Lachydrin©), beta hydroxyacid products (including salicylic acid), poly hydroxyacid products, retinol products, acetyl glucosamine or other effective anti-aging topical products on the face 2 weeks prior to the start of the study and throughout the duration of the study.
7. Completion and signing of a Informed Consent and Enrollment form, HIPAA form, photo release form, medical intake, skin habits survey.
8. Willingness to complete all study assessments.

   -

Exclusion Criteria:

1. Individuals who currently or in the last month have regularly used certain topical or oral medications which, in the opinion of the Investigators, may interfere with the study or that may expose study participants to unacceptable risks. Such products include oral prescription steroids or anti-inflammatories, topical steroids, or prescription skin treatment except for mild acne, as determined by the investigators.
2. Subjects who have a history of disease or current disease or regularly use topical or oral medications which, in the opinion of the Investigator, may interfere with the study or that may expose study participants to unacceptable risks. (i.e. oral or topical steroids or anti-inflammatories, etc.).
3. Uncontrolled metabolic disease such as diabetes, hyperthyroidism, or hypothyroidism or active Hepatitis, immune deficiency, or autoimmune disease as determined by the health questionnaire.
4. Pregnancy, nursing, or planning to become pregnant during the course of the study as determined by the health questionnaire.
5. History of skin cancer within the past 6 months.
6. Use of topical prescription retinoids for anti-aging including Retin-A®, Retin-A Micro®, Renova®, Avita®, Tazorac®, or Differin® within 2 weeks prior to the start of the study.

   Use of oral retinoids within 6 months of the study start.
7. Subjects must not have had mid-depth or superficial chemical peel or other anti-aging procedures on the face (laser, intense pulsed light, injectable fillers microdermabrasion, etc.) within 2 months of the study start.
8. Known allergies or sensitivities to test material ingredients or any topical skin care product (i.e., alpha hydroxyacids, retinol, sunscreens, moisturizers, cleansers, masques, toners, etc.).
9. Individuals currently participating in other clinical testing.
10. Start of hormone use (including for birth control) or changed hormones less than three months prior to the start of the study. Qualified subjects must not be taking hormones or must have been taking them for at least three months prior to the study start.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Genetic Profile & Product Response | 6 weeks
  The primary endpoint being studied in this study is the association of the product response to the 17 candidate SNP genotypes.

SECONDARY OUTCOMES:
Novel SNP Identification | 6 weeks
  The secondary endpoint will be identification of novel SNPs through genome-wide association analysis that may be associated with response to the study product.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Lee, MD, MA, Principal Investigator — Member
Locations (1):
- Halcyon Dermatology, Laguna Hills, California, United States

IPD SHARING:
Plan to Share IPD: No